CLINICAL TRIAL: NCT00576043
Title: Effect of Virtual Endoscopy Simulator Training on Real Patient Endoscopy: A Randomized, Controlled Trial
Brief Title: Effect of Virtual Endoscopy Simulator Training on Real Patient Endoscopy
Acronym: endosim
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Arnulf Ferlitsch, MD, Gastroenterology and Hepatology, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: endosim
Record Dates: First submitted 2007-12-17; First posted 2007-12-18 (Estimated); Last update posted 2008-03-27 (Estimated); Status verified 2008-03

CONDITIONS: Pain
Keywords: training; Patient satisfaction; endoscopy; simulator; Safety
MeSH Terms: conditions — Pain; Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: Training (Active Comparator): 3 weeks/2 hours per day of structured training for a total of 20 hours on the virtual endoscopy simulator
  Interventions: Procedure: Simulator Training
- 2: No Training (No Intervention): No simulator training before starting endoscopy training on real patients

INTERVENTIONS:
Procedure: Simulator Training — 3 weeks/2 hours per day of structured training for a total of 20 hours on the virtual endoscopy simulator with the GI-Mentor Virtual simulator device
  Arms: 1: Training

SUMMARY:
Trainees (Residents in internal medicine), naive to real patient endoscopy, will be randomized to receive either 3 weeks/2 hours per day of structured training for a total of 20 hours on the virtual endoscopy simulator GI-Mentor or no training before starting on-patient endoscopy in the University of Vienna Medical School Endoscopy Unit. Patients satisfaction and pain, technical accuracy and number of found/missed pathologies as well as average time for successful endoscopy will be recorded. After one month or 50 supervised, self performed endoscopies, trainees will be evaluated again with the above mentioned criteria during ten consecutive investigations.

ELIGIBILITY:
Inclusion Criteria:

* Trainees: naive to real patient endoscopy before training phase

Exclusion Criteria:

* Medical doctors with experience in gastrointestinal endoscopy
* Patients sedated for upper GI endoscopy
* Patients unwilling or unable to sign informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2004-03; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction measured on a visual analogue scale (VAS) | once immediately after patient endoscopy

SECONDARY OUTCOMES:
pain during endoscopy, measured with patient documentation on a visual analogue scale (VAS) | once immediately after patient endoscopy
technical accuracy (oral introduction of the scope into the esophagus, ability of passing the endoscope through the pylorus, inversion of the scope in the gastric fundus) | during endoscopy
number of found/missed pathologies | during endoscopy
average time for successful endoscopy | during endoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Arnulf Ferlitsch, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Internal Medicine III, Div. of Gastroenterology and Hepatology, Endoscopy Unit, Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Background] Ferlitsch A, Glauninger P, Gupper A, Schillinger M, Haefner M, Gangl A, Schoefl R. Evaluation of a virtual endoscopy simulator for training in gastrointestinal endoscopy. Endoscopy. 2002 Sep;34(9):698-702. doi: 10.1055/s-2002-33456. PMID 12195326